CLINICAL TRIAL: NCT04659369
Title: Study of Pharmacokinetic, Safety, Immunogenicity and Efficacy of CMAB819 and Nivolumab in Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of Pharmacokinetic, Safety, Immunogenicity and Efficacy of CMAB819 and Nivolumab in R/M HNSCC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficult to recruit subjects
Sponsor: Taizhou Mabtech Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMAB819-001
Record Dates: First submitted 2020-11-19; First posted 2020-12-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-05

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CMAB819 (Experimental): CMAB819 480 mg intravenous (IV) solution for Injection every 4 weeks until documented disease progression, discontinuation, withdrawal of consent or the study ends.
  Interventions: Drug: CMAB819
- Nivolumab (Active Comparator): Nivolumab 480 mg intravenous (IV) solution for injection every 4 weeks until documented disease progression, discontinuation, withdrawal of consent, or the study ends or up to 4 doses in subjects without disease progression, whichever occurs earlier. After completing 4 doses of Nivolumab therapy, administer of CMAB819 480 mg intravenous (IV) solution for injection every 4 weeks until documented disease progression, discontinuation, withdrawal of consent or the study ends.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: CMAB819 — for injection only
  Arms: CMAB819
Drug: Nivolumab — for injection only
  Other Names: Opdivo
  Arms: Nivolumab

SUMMARY:
The purpose of this study is to compare the pharmacokinetic, safety, immunogenicity and efficacy of CMAB819 and Nivolumab in subjects with recurrent or metastatic head and neck squamous cell carcinoma., after failure of prior platinum-based chemotherapy.

DETAILED DESCRIPTION:
Patients were randomized to receive CMAB819 or Nivolumab 480 mg by intravenous infusion every 4 weeks until documented disease progression, discontinuation, withdrawal of consent, or up to 4 doses in subjects without disease progression, whichever occurs earlier. After completing 4 doses of therapy, administer of CMAB819 480 mg intravenous (IV) solution for injection every 4 weeks until documented disease progression, discontinuation, withdrawal of consent or the study ends. Randomization was stratified by Eastern Cooperative Oncology Group (ECOG) performance status ECOG (0 versus 1), sex (male versus female), weight （≤60 kg versus >60kg）and clinical trial institution (up to 20 centers) .

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, Aged ≥18 years and ≤75 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status of ≤1.
3. Life expectancy of at least 3 months.
4. Histologically or cytologically confirmed recurrent or metastatic SCCHN (oropharynx, oral cavity, hypopharynx, larynx, etc.), Stage III/IV and not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy).
5. Tumor tissue (archival or fresh biopsy specimen wthin 3 years) must be available for PD-L1 expression analysis.
6. Subjects must have experienced disease recurrence or progression during or after last dose of platinum therapy for advanced or metastatic disease.

   (i)Subjects who received adjuvant or neoadjuvant platinum-based chemotherapy (after surgery and/or radiation therapy) and developed recurrent or metastatic disease within 3~6 months of completing therapy are eligible. (ii)Subjects with recurrent disease > 6 months after adjuvant or neoadjuvant platinum-based chemotherapy, who also subsequently progressed during or after a platinum- doublet regimen given to treat the recurrence, are eligible.
7. Subjects must have measurable disease by CT or MRI per RECIST 1.1 criteria.
8. All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE version 5.0) or baseline before administration of study drug. Subjects with toxicities attributed to prior anti-cancer therapy which are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum based therapy, are permitted to enroll.
9. Medically accepted effective contraception if procreative potential exists (applicable for both male and female subjects until at least 6 months after the last dose of trial treatment).
10. All baseline laboratory requirements will be assessed and should be obtained within -14 days of randomization. Screening laboratory values must meet the following criteria： (i) Blood routine: (a) Neutrophils ≥ 1.5 x 10^9/L；(b) Platelets ≥ 75 x 10^9/L；(c) Hemoglobin ≥ 90 g/L.

    (ii) Liver function: (a) AST ≤ 1.5 x ULN (subjects with liver metastasis≤ 5 x ULN); (b) ALT ≤ 1.5 x ULN (subjects with liver metastasis≤ 5 x ULN); (c) Total bilirubin ≤ 1.5 ULN [except subjects with Gilbert Syndrome who must have total bilirubin < 2.5 x ULN（3.0 mg/dL)].

    (iii) Renal function: (a) Serum creatinine of ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/minute (using Cockcroft/Gault formula).
11. Signed the informed consent form voluntarily.

Exclusion Criteria:

1. Histologically or cytologically confirmed recurrent or metastatic nasopharyngeal darcinoma, squamous carcinoma of unknown primary, salivary gland carcinoma, or cutaneous squamous cell carcinoma.
2. Subjects with active CNS metastases and/or carcinomatous meningitis. Subjects are eligible if CNS metastases are adequately treated and subjects are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to enrollment. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent).
3. Subjects with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) within the previous 3 years are excluded unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required during the study period.
4. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
5. Subjects with immunodeficiency inculding testing positive for human immunodeficiency virus (HIV) , acquired or congenital immunodeficiency disease, or organ transplantation.
6. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 （such as ipilimumab）antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
7. Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
8. Subjects with significant cardiovascular or cerebrovascular disease, such as dysrhythmias, conduction block, QTc interval at rest > 480 ms, New York Heart Association cardiac disease Class II or greater, left ventricular ejection fraction (LVEF) <50％, uncontrollable high blood pressures, or the following within 6 months prior to the first dosing: acute coronary syndrome, congestive heart-failure, aoreic dissection, stroke or any other Grade 3 or 4 adverse events of cardia and cerebrovascular disorder.
9. Treatment with Radical radiotherapy within 4 weeks prior to randomization; Treatment with palliative radiotherapy and anticancer effects of chinese herbal medicine within 2 weeks prior to randomization.
10. Has not recovered from the effects of major surgery or significant traumatic injury within 4 weeks prior to randomization.
11. Treatment with any investigational agent or devices within 4 weeks prior to randomization.
12. Treatment with any live attenuated vaccine within 4 weeks prior to randomization; Treatment with transfusion, hemopoietin, granulocyte colony-stimulating factor (G-CSF) or granulocyte macrophage-colony stimulating factor within 2 weeks prior to randomization.
13. Antitumor therapy except for study treatment are already ongoing or planned.
14. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive/immunoenhanced medications within 2 weeks prior to randomization. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
15. Positive test for hepatitis B virus surface antigen (HBV sAg) and HBV-DNA ≥1×10^3 copies/mL; Positive test for hepatitis C virus antibody.
16. History of allergy or intolerance (unacceptable adverse event) to study drug components, Polysorbate-80-containing infusions or other monoclonal antibodies.
17. Subjects with any other serious or uncontrollable medical conditions, active infection, physical examination abnormality, laboratory examination abnormality, altered mental state or mental illness, which is believed by investigator may increase the risk to the subjects or affect the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
AUC0-4w,1 | Day 1 to Day 29
  Area under the concentration-time curve (AUC) from time of the first dosing to time of 672 hours after the end of infusion.

SECONDARY OUTCOMES:
Cmax1 | Day 1 to Day 29.
  Maximum serum concentration from time of the first dosing to time of 672 hours after the end of infusion.
Cmin1 | Day 1 to Day 29.
  Minimum serum concentration from time of the first dosing to time of 672 hours after the end of infusion.
Tmax1 | Day 1 to Day 29
  Time to maximum of blood concentration from time of the first dosing to time of 672 hours after the end of infusion.
AUC0-4w,4 | From time of the fouth dosing to time of 672 hours after the end of infusion.
  Area under the concentration-time curve (AUC) from time of the fourth dosing to time of 672 hours after the end of infusion .
Cmax4 | From time of the fourth dosing to time of 672 hours after the end of infusion.
  Maximum serum concentration from time of the fourth dosing to time of 672 hours after the end of infusion.
Cmin4 | From time of the fourth dosing to time of 672 hours after the end of infusion.
  Minimum serum concentration from time of the fourth dosing to time of 672 hours after the end of infusion.
Tmax4 | From time of the fourth dosing to time of 672 hours after the end of infusion.
  Time to maximum of blood concentration from time of the fourth dosing to time of 672 hours after the end of infusion.
Adverse event frequencies | Date of the first dosing of study drug to 28 days post last dose of study drug.
  Number of Participants With Death, Study Drug-Related Death, Serious Adverse Events (SAEs), Drug-Related AEs, Deaths, Discontinuation of Study Drug Due to AE, and Immune-related AEs (irAEs) in Safety Population
Incidence of anti-drug antibodies. | Date of first doing of study drug to 28 days post last dose of study drug.
  Incidence of anti-drug antibodies.
Incidence of neutralizing antibody | Date of first dosing of study drug to 28 days post last dose of study drug.
  Incidence of neutralizing antibody
ORR16w | Randomization to disease progression, study drug is discontinued or 16 weeks after the end of infusion of the first dosing, whichever occurs first
  ORR was defined as the proportion of randomized participants who achieved a best response of complete response (CR) or partial response (PR) using the RECIST1.1 criteria as per investigator assessment.
DCR16w | Randomization to disease progression, study drug is discontinued or 16 weeks after the end of infusion of the first dosing, whichever occurs first
  DCR was defined as the proportion of randomized participants who achieved a best response of complete response (CR) , partial response (PR) or stable disease (SD) ≥6 weeks using the RECIST1.1 criteria as per investigator assessment.
PFSR16w | Randomization to disease progression, study drug is discontinued or 16 weeks after the end of infusion of the first dosing, whichever occurs first.
  PFS was defined as the time between the date of randomization and the first date of documented progression, as determined by the investigator (as per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria), or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Ph.D, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China